CLINICAL TRIAL: NCT03908047
Title: Feasibility of Detecting Functional Changes in the Brain After Tibial Nerve Stimulation and the Association with the Sacral Roots Architecture: a Pilot Magnetic Resonance Study
Brief Title: Functional Changes in the Brain After Tibial Nerve Stimulation: a Pilot Study
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2019-01
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injuries; Bladder, Neurogenic
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- healthy volunteers
  Interventions: Other: magnetic resonance imaging

INTERVENTIONS:
Other: magnetic resonance imaging — functional magnetic resonance imaging and diffusion tensor imaging after tibialis nerve stimulation

SUMMARY:
The lower urinary tract is innervated by the autonomous (sympathetic, parasympathetic) and the somatic nervous system. Afferent information from the lower urinary tract (LUT) (e.g. filling state and volume of the urinary bladder) is conducted via the dorsal roots to the sacral spinal cord and from there to the pontine micturition center (PMC) in the brain stem. The PMC has several connections to other cortical areas. These complex interactions with the cortex enable voluntary control of the LUT and are crucial for urinary continence. The integrity of this neuronal circuit is crucial for an undisturbed function. Deterioration of the nerve fibers due to a systemic neurological disease (e.g. spinal cord injury) can affect LUT function. Neurogenic lower urinary tract dysfunction can lead to urgency, urge incontinence, reduced bladder capacity and secondary deterioration of the upper urinary tract (i.e. kidneys). First-line therapy of neurogenic detrusor overactivity contains antimuscarinic treatment. In case of side effects or remaining detrusor overactivity, nerve stimulation (e.g. sacral neuromodulation and in effect nerve tibialis stimulation) is an accepted therapy option. The precise mechanism of action of these neuro-modulatory procedures is still unknown. Utilizing state-of-the-art neuroimaging techniques, we intend to investigate the functional activation pattern after afferent tibialis nerve stimulation as well as the association with the architecture of the sacral roots. We aime to get a better insight into functional neuromodulation and central nervous processing. The study aim is to evaluate the feasibility in healthy subjects as a pilot study for the application of these method in patients with chronic, incomplete spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* 18-50 years old
* informed consent

Exclusion Criteria:

* history of neurological disease (eg. multiple sclerosis, epilepsy)
* cardiac pacemaker, insulin or other pumps
* claustrophobia
* pathological findings in the uroflowmetry or post void residual assessment
* medication with central nervous effects
* pregnancy or lactating
* unable to give informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
change in functional network connectivity | baseline; 30 minutes during nerve stimulation
  change in brain network activity identified by independent component analysis

OTHER OUTCOMES:
gender | baseline
  male or female
age | baseline
  time since birth in years

CONTACTS AND LOCATIONS:
Overall Officials: Jens Wöllner, Dr., Principal Investigator — Senior Consultant Neuro-Urology
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No